CLINICAL TRIAL: NCT01771965
Title: Increasing Treatment Seeking Among Suicidal Veterans Calling the Crisis Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 11-298
Record Dates: First submitted 2012-12-21; First posted 2013-01-18 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): No intervention.
- CB Intervention (Experimental): Cognitive Behavioral one-on-one single session administered by phone
  Interventions: Behavioral: CB Intervention

INTERVENTIONS:
Behavioral: CB Intervention — The Cognitive Behavioral (CB) intervention is a brief, manualized, tailored one-on-one single session lasting 45-60 minutes and administered by phone. An individual format was chosen to reduce the potential discomfort of stigma of individual concerns in the presence of others. The intervention targets a change in the beliefs that influence whether or not someone enters mental health or substance use treatment. During the session, participants will be given a brief introduction to CBT and informed that CBT is based on the theory that cognitions (i.e., thoughts/beliefs), feelings and behaviors all interact with each other;101, 102 therefore, thoughts about certain situations or things influence behavior. Since thoughts are modifiable, changing thoughts about situations may change behavior.
  Arms: CB Intervention

SUMMARY:
The goal of this research plan is to test the effectiveness of a brief, cognitive behavioral (CB) intervention to promote behavioral health treatment engagement among at-risk Veterans who call the Crisis Line but are resistant to behavioral health services.

DETAILED DESCRIPTION:
The goal of this research plan is to test the effectiveness of a brief, cognitive behavioral (CB) intervention to promote behavioral health treatment engagement among at-risk Veterans who call the Crisis Line but are resistant to behavioral health services. This randomized controlled trial will recruit 80 Veterans who report current suicidal ideation at the time of the Crisis Line call and are resistant to seeking behavioral health treatment. Half of the participants will receive the brief, individualized CB intervention and half will receive standardized procedures from VA's Crisis Line (i.e., usual care). The effectiveness of the intervention will be tested on 1) attitudes toward behavioral health treatment rates, and 2) initiation of and adherence to treatment (assessed by the number of sessions attended). The investigators will also assess the impact of the intervention on suicidal ideation (SI) and explore the impact on the most common symptoms observed in Veteran suicide decedents (e.g., depression).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the study are as follows:

* individuals 18 and older who call the Veteran Crisis Line
* have a phone number where they can be reached, be it a land line or a cell phone
* deemed by the Crisis Line responder to be at risk for suicide, but not imminent risk
* refuse a referral to the SPC or to a behavioral health treatment provider during the call
* report current suicidal ideation (SI) during the call based on administration of a standard item
* have not been in behavioral health treatment in the past. Presence of SI will be subsequently confirmed by the research assistant using the Columbia Suicide Severity Rating Scale, a validated instrument.

Exclusion Criteria:

Exclusion criteria are being judged by the Crisis Line responder to show:

* debilitating cognitive impairment
* active psychosis or mania
* acute alcohol or drug intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A. Stecker, PhD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (2):
- United States (2):
  - Canandaigua VA Medical Center, Canandaigua, NY, Canandaigua, New York
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial implemented the intervention at the VA's National Crisis Line during a period of dynamic change at the Crisis Line including turnover of top leadership and major changes in procedures and personnel.
  Our bottom line recruitment numbers were low.
Period: Overall Study
Arm/Group | Usual Care | CB Intervention
Started | 10 | 9
Completed | 7 | 4
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | CB Intervention | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (17.9) | 39.8 (14.6) | 41.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Treatment Engagement (Number of Participants Entering Treatment)
Description: The investigators will be asking about service utilization since baseline interview. Zero = no mental health treatment and 1 = received mental health treatment.
Time Frame: 30 days after baseline
Population: Only 7 of the 10 control participants and 4 of the 9 intervention participants completed follow-up assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | CB Intervention
Number analyzed (Participants) | 7 | 4
Participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Usual Care | CB Intervention
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No